CLINICAL TRIAL: NCT04757272
Title: Does Hepatitis C Management Protect Egyptian Population Against Severe Corona Virus Disease-2019 (COVID-19)?
Brief Title: Does Hepatitis C Management Protect Egyptian Population Against Severe Corona Virus Disease-2019?
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Sherif M. S. Mowafy, Associate professor of anesthesia and surgical intensive care, Zagazig University
Other Study IDs: 6733-24-2-2021
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Corona Virus Infection; Hepatitis
MeSH Terms: conditions — Coronavirus Infections; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Modulation of the renin angiotensin system by the chronic hepatitis C virus treatment either by (Daclatasvir and Sofosbuvir), (Daclatasvir and Sofosbuvir plus Ribavirin), or (Ribavirin and Interferon) protocols could give an explanation for the low incidence of COVID-19 among Egyptian population. Adding it may play a role in COVID 19 prophylaxis.

DETAILED DESCRIPTION:
The interaction of severe acute respiratory syndrome corona virus-2 (SARS-CoV-2) and the renin angiotensin system (RAS) via angiotensin converting enzyme-2 (ACE-2), the receptor used by the SARS-CoV-2 to gain access to cells could provide an explanation for the several unusual clinical findings observed in COVID-19 Although chronic hepatitis is one of the risk factors listed by WHO for severe COVID-19, low incidence of COVID-19 was observed among HCV patients admitted to Egyptian hospitals.

Modulation of the RAS by the chronic hepatitis C virus treatment either by (ACEI or ARBS), (Daclatasvir and Sofosbuvir), (Daclatasvir and Sofosbuvir plus Ribavirin), or (Ribavirin and Interferon) protocols could give an explanation for the low incidence of COVID-19 among Egyptian population. Adding it may play a role in COVID 19 prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients who were diagnosed to have COVID-19 and admitted to Zagazig University Hospitals during the period from May 2020 to January 2021

Exclusion Criteria:

-

Ages: 21 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who were diagnosed to have COVID-19 during the period from May 2020 to march 2022 were included and their medical records were analyzed for the previous history of chronic hepatitis C and its management protocols. Any history to receive HCV treatment either (ACEI or ARBS), (Daclatasvir and Sofosbuvir), (Daclatasvir and Sofosbuvir plus Ribavirin), or (Ribavirin and Interferon) management protocols will be recorded
Sampling Method: Probability Sample
Enrollment: 2106 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
incidence of chronic hepatitis C among COVID-19 hospitalized patients. | 7 months
  incidence of chronic hepatitis C among COVID-19 hospitalized patients.

SECONDARY OUTCOMES:
the impact of previous exposure to different HCV management protocols on the clinical characteristics and outcome of COVID-19 among COVID-19 hospitalized patients | 7 months
  the impact of previous exposure to different HCV management protocols on the clinical characteristics and outcome of COVID-19 among COVID-19 hospitalized patients

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication
Access Criteria: by contacting the principal investigator

REFERENCES:
- [Background] Wiese OJ, Allwood BW, Zemlin AE. COVID-19 and the renin-angiotensin system (RAS): A spark that sets the forest alight? Med Hypotheses. 2020 Nov;144:110231. doi: 10.1016/j.mehy.2020.110231. Epub 2020 Sep 3. PMID 33254538
- [Background] Paz Ocaranza M, Riquelme JA, Garcia L, Jalil JE, Chiong M, Santos RAS, Lavandero S. Counter-regulatory renin-angiotensin system in cardiovascular disease. Nat Rev Cardiol. 2020 Feb;17(2):116-129. doi: 10.1038/s41569-019-0244-8. Epub 2019 Aug 19. PMID 31427727
- [Background] Imai Y, Kuba K, Rao S, Huan Y, Guo F, Guan B, Yang P, Sarao R, Wada T, Leong-Poi H, Crackower MA, Fukamizu A, Hui CC, Hein L, Uhlig S, Slutsky AS, Jiang C, Penninger JM. Angiotensin-converting enzyme 2 protects from severe acute lung failure. Nature. 2005 Jul 7;436(7047):112-6. doi: 10.1038/nature03712. PMID 16001071
- [Background] Li W, Moore MJ, Vasilieva N, Sui J, Wong SK, Berne MA, Somasundaran M, Sullivan JL, Luzuriaga K, Greenough TC, Choe H, Farzan M. Angiotensin-converting enzyme 2 is a functional receptor for the SARS coronavirus. Nature. 2003 Nov 27;426(6965):450-4. doi: 10.1038/nature02145. PMID 14647384
- [Background] Husic-Selimovic A, Sofic A, Huskic J, Bulja D. Effect of Antiviral Therapy on Serum Activity of Angiotensin Converting Enzyme in Patients with Chronic Hepatitis C. Med Arch. 2016 Apr;70(2):92-6. doi: 10.5455/medarh.2016.70.92-96. Epub 2016 Apr 1. PMID 27147779
- [Background] Zakaria S, El-Sisi AE. Daclatasvir and Sofosbuvir Mitigate Hepatic Fibrosis Through Downregulation of TNF-alpha / NF-kappaB Signaling Pathway. Curr Mol Pharmacol. 2020;13(4):318-327. doi: 10.2174/1874467213666200116114919. PMID 31951178
- [Background] Omran D, Alboraie M, Zayed RA, Wifi MN, Naguib M, Eltabbakh M, Abdellah M, Sherief AF, Maklad S, Eldemellawy HH, Saad OK, Khamiss DM, El Kassas M. Towards hepatitis C virus elimination: Egyptian experience, achievements and limitations. World J Gastroenterol. 2018 Oct 14;24(38):4330-4340. doi: 10.3748/wjg.v24.i38.4330. PMID 30344418
- [Background] Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW; the Northwell COVID-19 Research Consortium; Barnaby DP, Becker LB, Chelico JD, Cohen SL, Cookingham J, Coppa K, Diefenbach MA, Dominello AJ, Duer-Hefele J, Falzon L, Gitlin J, Hajizadeh N, Harvin TG, Hirschwerk DA, Kim EJ, Kozel ZM, Marrast LM, Mogavero JN, Osorio GA, Qiu M, Zanos TP. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. JAMA. 2020 May 26;323(20):2052-2059. doi: 10.1001/jama.2020.6775. PMID 32320003